CLINICAL TRIAL: NCT00819026
Title: Observational Trial of Hepatitis C Virus Infected Patients on Calcineurin Inhibitors
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: UWisHCV-1
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — viral RNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Hepatitis C Virus is constantly evolving genetically, particularly in response to the immune system. This is an observational study to examine if immunosuppressants particularly calcineurin inhibitors taken by transplant patients in order to avoid organ rejection causes predictable changes in the genetics of this virus that might be important in order to treat it effectively.

ELIGIBILITY:
Inclusion Criteria:

* HCV infected on immunosuppression

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: solid organ transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2008-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Striker, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Result] Ansari IU, Allen T, Berical A, Stock PG, Barin B, Striker R. Phenotypic analysis of NS5A variant from liver transplant patient with increased cyclosporine susceptibility. Virology. 2013 Feb 20;436(2):268-73. doi: 10.1016/j.virol.2012.11.018. Epub 2013 Jan 2. PMID 23290631